

Investigative Medicine 6<sup>th</sup> floor, Commonwealth Building Imperial College Faculty of Medicine Hammersmith Hospital Du Cane Road London W12 ONN

London - Queen Square REC Ref 18/LO/0376 IRAS ID 236553 Version 4.0 14/01/2020

## **Participant Consent Form**

Title of project:

## Investigating physiological effects of weight loss on male fertility

| The participant should complete the whole of this sheet himself. |
|---|
| (please initial each statement if it applies to you) |
| The study has been explained to me by: Prof/Dr/Mr/Mrs/Ms |
| I have read the Information Sheet for research participants (versiondate). I was given the opportunity to ask questions and discuss this study. I received satisfactory answers to all my questions, and received enough information about the study. |
| I understand that I am free to withdraw from the study at any time, without having to give a reason for withdrawing and without affecting my future medical care. |
| I understand NHS clinicians working on this research study who are not part of the usual care team will have access to medical records. Also authorised persons from the sponsor, NHS and regulatory authorities may have access to my medical records. |
| I agree for my blood and semen to be taken to find more about the effects of weight loss on male infertility. |
| My personal details may be stored on password protected Imperial College Healthcare NHS Trust computers for the purpose of this study. This information will be kept strictly confidential. Data will be stored for 10 years according to Imperial College Data Management policy. Processing of personal details will follow the principles as set out in the Data Protection Act 1998. |
| Identifiable data (e.g. consent forms) may be kept in a locked office within Imperial College London or Imperial College Healthcare NHS Trust. Data will be stored for 10 years according to Imperial College Data Management policy. |
| If I can no longer make decisions (lose capacity) during the study, then I will be withdrawn from the study but agree that any data or results already collected can be used in the study. |
| I agree to take part in this study. |
| I agree for my GP to be notified that I took part in the study via a standard letter |
| SignedDate |
| (NAME IN BLOCK CAPITALS) |
| Investigator's signature |
| (NAME IN BLOCK CAPITALS) |